CLINICAL TRIAL: NCT02964975
Title: Quality of Life Assessment in Patients With Coronary Artery Chronic Total Occlusion: Randomized Comparison of Optimal Medical Therapy and Percutaneous Coronary Intervention
Brief Title: Randomized Comparison of Optimal Medical Therapy and Percutaneous Recanalization for Chronic Total Occlusion (COMET-CTO)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Sinisa Stojkovic, Head Deaprtment of Interventional Cardiologyand Catheter Ablation, Principal Investigator, Clinical Professor, Clinical Centre of Serbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBVSS-30
Record Dates: First submitted 2016-11-13; First posted 2016-11-16 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Chronic Total Occlusions of Coronary Arteries
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optimal medical therapy (Active Comparator): conservative treatment
  Interventions: Drug: Optimal medical therapy
- Percutaneous coronary intervention (Active Comparator): Percutaneous coronary intervention of chronic total occlusion
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Recanalisation of chronic total occlusion of coronary artery
  Other Names: PCI
  Arms: Percutaneous coronary intervention
Drug: Optimal medical therapy — Medical threatment according to guidelines
  Other Names: Angina pectoris opetimal medical therapy
  Arms: Optimal medical therapy

SUMMARY:
Several meta analysis comparing successful Percutaneous Coronary Intervention of Chronic Total Occlusion (PCI-CTO) with unsuccessful PCI-CTO showed that there is significant reduction in short-term and long-term mortality. To our knowledge till today no prospective randomized trial compared percutaneous revascularization of CTO with optimal medical therapy. For this reason quality of live improvement is one of the most important indications for revascularization in elective patients with CTO. In contemporary literature Seattle Angina Questionnaire (SAQ) is a psychometrically solid disease-specific instrument designed to assess the functional status of patients with angina. It comprises 19 questions that quantify five clinically relevant domains: physical limitation, angina stability, angina frequency, treatment satisfaction and disease perception/quality of life.

In this open prospective study patients with CTO of coronary artery will be randomized in two groups: first - patients with percutaneous coronary intervention of chronic total occlusion with optimal medical therapy and second group - patients with only optimal medical therapy (control group). Primary endpoint will be quality of life and secondary endpoints will be mayor adverse cardiovascular events (MACE). All patients will complete Seattle Angina Questionnaire before randomization and after 6 months of follow-up.

DETAILED DESCRIPTION:
Coronary artery chronic total occlusion (CTO) is defined as complete occlusion of coronary arteries that lasts for more than three months (TIMI 0 coronary flow in occluded segment). In absence of serial angiograms , occlusion duration can be assumed based on clinical data regarding event that caused occlusion. Consensus document from the Euro CTO club suggests 3 levels of certainty:

a) Certain (angiographically confirmed): the minority of cases where a previous angiogram (for instance before a previous CABG operation, or after an acute myocardial infarction) has confirmed the presence of TIMI 0 flow for > 3 months prior to the planned procedure; b) Likely (clinically confirmed): objective evidence of an acute myocardial infarction in the territory of the occluded artery without other possible culprit arteries >3 months before the current angiogram; c) Possible (undetermined): a CTO with TIMI 0 flow and angiographic anatomy suggestive of long-standing occlusion (collateral development, no contrast staining) with stable angina symptoms unchanged in the last 3 months or evidence of silent ischemia; in case of recent acute ischemic episodes (acute myocardial infarction or unstable angina or worsening effort angina), a culprit artery other than the occluded vessel should be present.

CTO is an often finding. In spite of that, there is uncertainty should this lesions be revascularized and in what way. If there are symptoms or objective proof of ischemia and viability in the area of occluded artery distribution, recanalization of CTO should be considered. Several studies showed that in the presence of chronic total occlusion collateral circulation may produce supply of oxygen and preserve viability. However assessment of collateral circulation with adenosine stress test showed abnormal coronary reserve in over than 90% was reduced which means that collaterals are not enough Therapeutically uncertainties lead partially from technical complex procedures of revascularization CTO with PCI, with success rate of 60-70% which is importantly lower than revascularization rate of non-CTO lesions (98%). During last decade there has been significant improvement in technology, equipment and techniques of percutaneous revascularization procedures for CTO that increased procedural success rate (around 90%). On the other hand there are separate views regarding possibility of treating this patients with coronary artery bypass graft (CABG), and specially patients with single coronary disease Metaanalysis performed by O'Connor SA et al. showed that presence of chronic total occlusion on non infarct artery in patients with acute myocardial infarction significantly increases mortality. Furthermore several mataanalyses that analyzed the effect of PCI CTO on survival, showed significant reduction of mortality rate in short term and also long term follow up. Studies enrolled in this metaanalyses were retrospective or prospective registries which compared successful PCI CTO with PCI CTO failure.

There are different explanations for this clinical result (mortality reduction):

1. direct benefit of achieving coronary flow and myocardial perfusion improves ventricular function and reduces risk of malignant arrhythmias
2. patients in which PCI was unsuccessful probably have more serious coronary atherosclerosis and fibrosis that contribute to procedural failure and greater mortality (3).

Similar to previous metaanalyses study conducted by Prasada et al. showed significantly greater mortality in the group with procedural failure .

Study conducted by Hoye et al. showed significant increase of 5-year mortality rate, CABG and MACE in the group with procedural failure. Authors explained the difference in survival by pharmacological management that can be confounding factor. Also authors stated that better prognosis after successful procedure is probably related to improved left ventricular function and reduced risk of malignant arrhythmias. To our knowledge, there is no prospective randomized study which compared PCI CTO with optimal medical therapy. For this reason quality of life improvement is one of the most important indication for revascularization CTO in elected patients. However, in contemporary literature there is little data regarding quality of life assessment in patients with CTO.

Quality of life assessment is important indicator of successful revascularization in patients with coronary artery disease. "Seattle Angina Questionnaire" (SAQ) is validated for quality of life assessment in patients with coronary artery disease. This questionnaire is based on five different domains : physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception. So far quality of life assessment with SAQ was used in four studies. Two of them compared results of SAQ in patients with successful recanalization of CTO and patients with procedural failure. They proved significant improvement in SAQ score in patients with recanalized CTO. Third study compared revascularization strategies (PCI vs. CABG) with optimal medical therapy in patients with diagnosed CTO. In the group treated with medical therapy there were no changes in scores of SAQ domains after one year follow-up, while in patients that were revascularized in CTO territory improvement in SAQ scores were documented in three domains (Physical restraint, angina frequency and disease perception). Fourth study compared quality of life after CTO PCI vs.PCI in on non CTO lesion. In both groups similar improvement was documented in all domains during 6 months follow-up.

So far no prospective randomized study was conducted that examined quality of life in patients with CTO.

ELIGIBILITY:
Inclusion Criteria:

* CTO of coronary artery (TIMI 0 flow)
* a) Stabile angina and/or b) evidence of ischemia in the territory of the CTO and/or c) evidence of viable myocardium in the CTO territory
* target coronary artery with a reference diameter of 2.5 mm

Exclusion Criteria:

* acute myocardial infarction in past month
* contraindications for dual antiplatelet therapy in future 12 months
* contraindications for drug eluting stents (DES)
* informed consent not signed
* CTO in bypass graft
* EF <20 %
* Dementia
* Patient not available for follow-up
* CVI or TIA in past 6 months
* Patients with:

  1. neutropenia (<1000 /mm3) in past two weeks
  2. thrombocytopenia (<100 000/mm3)
  3. AST, ALT, alkaline phosphatase >1.5x the upper limit of normal
  4. serum creatine >2 mg/dL (>180 µmol/L)
* Patients with allergy to iodine contrast that cannot be treated medically
* Life expectancy not longer than one year
* Patients with bleeding diathesis or coagulopathy or will refuse transfusions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | 6 months
  Seattle Angina Questionnaire

SECONDARY OUTCOMES:
all cause death, Major Adverse Cardiac Event (MACE) including: Acute Myocardial Infarction - AMI, repeated revascularisation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sinisa Stojkovic, PhD, Principal Investigator — Clinical Centre of Serbia
Locations (1):
- Clinical Centre os Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sianos G, Werner GS, Galassi AR, Papafaklis MI, Escaned J, Hildick-Smith D, Christiansen EH, Gershlick A, Carlino M, Karlas A, Konstantinidis NV, Tomasello SD, Di Mario C, Reifart N; EuroCTO Club. Recanalisation of chronic total coronary occlusions: 2012 consensus document from the EuroCTO club. EuroIntervention. 2012 May 15;8(1):139-45. doi: 10.4244/EIJV8I1A21. No abstract available. PMID 22580257
- [Background] Fefer P, Knudtson ML, Cheema AN, Galbraith PD, Osherov AB, Yalonetsky S, Gannot S, Samuel M, Weisbrod M, Bierstone D, Sparkes JD, Wright GA, Strauss BH. Current perspectives on coronary chronic total occlusions: the Canadian Multicenter Chronic Total Occlusions Registry. J Am Coll Cardiol. 2012 Mar 13;59(11):991-7. doi: 10.1016/j.jacc.2011.12.007. PMID 22402070
- [Background] Prasad A, Rihal CS, Lennon RJ, Wiste HJ, Singh M, Holmes DR Jr. Trends in outcomes after percutaneous coronary intervention for chronic total occlusions: a 25-year experience from the Mayo Clinic. J Am Coll Cardiol. 2007 Apr 17;49(15):1611-1618. doi: 10.1016/j.jacc.2006.12.040. Epub 2007 Apr 2. PMID 17433951
- [Background] Werner GS, Bahrmann P, Mutschke O, Emig U, Betge S, Ferrari M, Figulla HR. Determinants of target vessel failure in chronic total coronary occlusions after stent implantation. The influence of collateral function and coronary hemodynamics. J Am Coll Cardiol. 2003 Jul 16;42(2):219-25. doi: 10.1016/s0735-1097(03)00624-7. PMID 12875755
- [Background] Rathore S, Matsuo H, Terashima M, Kinoshita Y, Kimura M, Tsuchikane E, Nasu K, Ehara M, Asakura Y, Katoh O, Suzuki T. Procedural and in-hospital outcomes after percutaneous coronary intervention for chronic total occlusions of coronary arteries 2002 to 2008: impact of novel guidewire techniques. JACC Cardiovasc Interv. 2009 Jun;2(6):489-97. doi: 10.1016/j.jcin.2009.04.008. PMID 19539251
- [Background] Saito S. Progress in angioplasty for chronic total occlusions again. Catheter Cardiovasc Interv. 2010 Nov 15;76(6):850-1. doi: 10.1002/ccd.22847. No abstract available. PMID 21104774
- [Background] Godino C, Sharp AS, Carlino M, Colombo A. Crossing CTOs-the tips, tricks, and specialist kit that can mean the difference between success and failure. Catheter Cardiovasc Interv. 2009 Dec 1;74(7):1019-46. doi: 10.1002/ccd.22161. PMID 19950136
- [Background] Maron DJ, Boden WE, O'Rourke RA, Hartigan PM, Calfas KJ, Mancini GB, Spertus JA, Dada M, Kostuk WJ, Knudtson M, Harris CL, Sedlis SP, Zoble RG, Title LM, Gosselin G, Nawaz S, Gau GT, Blaustein AS, Bates ER, Shaw LJ, Berman DS, Chaitman BR, Weintraub WS, Teo KK; COURAGE Trial Research Group. Intensive multifactorial intervention for stable coronary artery disease: optimal medical therapy in the COURAGE (Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation) trial. J Am Coll Cardiol. 2010 Mar 30;55(13):1348-58. doi: 10.1016/j.jacc.2009.10.062. PMID 20338496
- [Background] Pancholy SB, Boruah P, Ahmed I, Kwan T, Patel TM, Saito S. Meta-analysis of effect on mortality of percutaneous recanalization of coronary chronic total occlusions using a stent-based strategy. Am J Cardiol. 2013 Feb 15;111(4):521-5. doi: 10.1016/j.amjcard.2012.10.034. PMID 23375252